CLINICAL TRIAL: NCT03512990
Title: Clinical And Anatomic Study Of An Ultrasound-Guided Selective Block Of The Superior Trunk Of The Brachial Plexus. Description Of A New Approach
Brief Title: Clinical And Anatomic Study Of An Ultrasound-Guided Superior Trunk Of The Brachial Plexus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, Professor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Superior Trunk
Record Dates: First submitted 2018-04-10; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Brachial Plexus Block; Shoulder Surgery
Keywords: Brachial Plexus Block; Superior Trunk; Phrenic Nerve

STUDY DESIGN:
Intervention Model Description: We suggest an injection more distally, where superior trunk is in costoclavicular space below omohyoid muscle, proximal to the suprascapular outlet. The needle is advanced below the prevertebral layer of deep cervical fascia, avoiding that the tip of the needle lies in the fascial plane between investing layer of deep vertebral fascia and prevertebral layer.
  Patients scheduled for rotator cuff surgery will receive 6 mL of 0,5% bupivacaine. Successful block is defined as motor score of ≤ 2 on modified Bromage scale in the deltoid and bíceps; absent sensation to cold and pinprick sensation in C5 and C6 dermatomes within 30 minutes of injection.
  To evaluate phrenic nerve, diaphragmatic excursion will be assessed by ultrasonography of ipsilateral hemidiaphragm and with impedance tomography.
  Moreover, 6 mL of methylene blue will be injected into cadavers to evaluate if dispersion was restricted to fibers of the superior trunk and don't reach phrenic nerve.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bupivacaine - Superior Trunk Block (Experimental): Patients scheduled for rotator cuff surgery received 6 mL of 0,5% bupivacaine in the superior Trunk.
  6 mL of methylene blue will be injected into cadavers with the same technique.
  Interventions: Procedure: Bupivacaine - Superior Trunk Block

INTERVENTIONS:
Procedure: Bupivacaine - Superior Trunk Block — It will be performed the superior trunk approach with local anesthestic in patients and methylene blue in cadavers.

SUMMARY:
Introduction

Interscalene brachial plexus block is the most commonly performed regional anesthesia technique to promote analgesia for shoulder surgeries. However, one of limitations is the risk of phrenic nerve palsy despite injection of low volumes, being contraindicated in patients with limited pulmonary reserve.

Burckett-St.Laurent et al described an alternative approach to avoid phrenic block - the superior trunk approach.

In this case series, the investigators suggest a modification of Burckett-St.Laurent's technique. The objective of this study is to evaluate efficacy, phrenic nerve function and contrast dispersion in cadavers after performing this new approach.

Materials and methods

The study was approved by Institutional Review Board of our institution. To perform the superior trunk approach described by Burckett-St.Laurent, C5 and C6 nerve roots are identified within the interscalene groove and traced distally to where they coalesce into the superior trunk, proximal to the takeoff of the suprascapular nerve. Burckett-St.Laurent et al suggest spreading local anesthetic around superior trunk at this point.

The investigators suggest an injection more distally, where superior trunk is in costoclavicular space below omohyoid muscle, proximal to the suprascapular outlet. The needle is advanced below the prevertebral layer of deep cervical fascia, avoiding that the tip of the needle lies in the fascial plane between investing layer of deep vertebral fascia and prevertebral layer, a loose fascial plane where lymph node chain is located and may allow postero-anterior dispersion toward phrenic. To guarentee right position of the tip the investigators suggest an intracluster pattern of spread.

Patients scheduled for rotator cuff surgery will receive 6 mL of 0,5% bupivacaine in this new approach. Successful block is defined as motor score of ≤ 2 on modified Bromage scale in the deltoid and bíceps; absent sensation to cold and pinprick sensation in C5 and C6 dermatomes within 30 minutes of injection.

To evaluate phrenic nerve, diaphragmatic excursion will be assessed by ultrasonography of ipsilateral hemidiaphragm and impedance tomography. Pain scores and analgesic consumption will be assessed in PACU.

Moreover, 6 mL of methylene blue will be injected into cadavers to evaluate if dispersion is restricted to fibers of the superior trunk and don't reach phrenic nerve.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* BMI < 35 kg/m²
* Patients scheduled for rotator cuff surgery

Exclusion Criteria:

* cognitive impairment or active psychiatric condition
* infection at the puncture site of the blockade
* coagulopathy
* history of allergy to bupivacaine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Superior Trunk Successful Block | within 30 minutes of injection
  Evaluate the efficacy of the block: Successful block was defined as motor score of ≤ 2 on modified Bromage scale in the deltoid and bíceps; absent sensation to cold and pinprick sensation in C5 and C6 dermatomes

SECONDARY OUTCOMES:
Phrenic nerve Block | at 30 minutes
  Evaluate the phrenic function after the block: To evaluate phrenic nerve, diaphragmatic excursion was assessed by ultrasonography of ipsilateral hemidiaphragm

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Franco CD, Williams JM. Ultrasound-Guided Interscalene Block: Reevaluation of the "Stoplight" Sign and Clinical Implications. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):452-9. doi: 10.1097/AAP.0000000000000407. PMID 27203394
- [Result] Burckett-St Laurent D, Chan V, Chin KJ. Refining the ultrasound-guided interscalene brachial plexus block: the superior trunk approach. Can J Anaesth. 2014 Dec;61(12):1098-102. doi: 10.1007/s12630-014-0237-3. Epub 2014 Sep 11. PMID 25208976
- [Result] Tran DQ, Elgueta MF, Aliste J, Finlayson RJ. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):32-38. doi: 10.1097/AAP.0000000000000529. PMID 27941477
- [Result] Franco CD. The Ultrasound Images of the Proximal Interscalene Space: A Reply to Dr Gabriel and Dr Sandhu. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):119-120. doi: 10.1097/AAP.0000000000000533. No abstract available. PMID 27997487
- [Result] Siegenthaler A, Moriggl B, Mlekusch S, Schliessbach J, Haug M, Curatolo M, Eichenberger U. Ultrasound-guided suprascapular nerve block, description of a novel supraclavicular approach. Reg Anesth Pain Med. 2012 May-Jun;37(3):325-8. doi: 10.1097/AAP.0b013e3182409168. PMID 22222688
- [Result] Wiegel M, Moriggl B, Schwarzkopf P, Petroff D, Reske AW. Anterior Suprascapular Nerve Block Versus Interscalene Brachial Plexus Block for Shoulder Surgery in the Outpatient Setting: A Randomized Controlled Patient- and Assessor-Blinded Trial. Reg Anesth Pain Med. 2017 May/Jun;42(3):310-318. doi: 10.1097/AAP.0000000000000573. PMID 28257388